CLINICAL TRIAL: NCT02039934
Title: Effect of High-intensity Low-volume Training on Insulin Sensitivity in Patients With Type 2 Diabetes and Healthy Lean Subjects
Brief Title: Effect of High-intensity Low-volume Training on Insulin Sensitivity in Type 2 Diabetes
Acronym: HIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: German Diabetes Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HIT and insulin sensitivity
Record Dates: First submitted 2012-09-07; First posted 2014-01-20 (Estimated); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Type 2 Diabetes
Keywords: type 2 diabetes; exercise intervention; high intensity interval training
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- high intensity interval training (Experimental): 30 minute sessions of high-intensity interval training on a bicycle ergometer three times per week
  Interventions: Other: High intensity interval training

INTERVENTIONS:
Other: High intensity interval training — The intervention consists of 30 minute sessions of high-intensity interval training on a bicycle ergometer three times per week.
  Training program: After 5 minutes of warm-up the subject cycles for 10 intervals of 60 s. at 90 % maximum effort separated 60 s at 20% maximum effort, based on a previously performed spiroergometry, followed by 5 minutes of cool-down.

SUMMARY:
High intensity interval training is applied for several diseases.

Hypothesis: High intensity interval training improves insulin sensitivity in patients with type 2 diabetes.

DETAILED DESCRIPTION:
Type 2 diabetes mellitus is a multifactorial metabolic disease that is characterized by reduced insulin sensitivity and insulin production leading to impaired glucose tolerance. Overweight and low physical activity are the main risk factors for the development of type 2 diabetes. Increased physical activity has shown to improve insulin sensitivity, hence, exercise plays a significant role in the prevention and therapy of type 2 diabetes. This study aims at investigating the acute and chronic effects of high-intensity low-volume training, that consists of brief bursts of very vigorous exercise separated by recovery periods, on metabolic function in patients with type 2 diabetes, people at high risk for the disease and healthy, lean individuals. Study participants take part in 30 min training session three times a week for a period of 12 weeks. Participants are studied on four occasions, prior to the intervention, after an acute bout of exercise as well as after 6 and 12 weeks of training in order to assess physical fitness, body composition, insulin sensitivity, energy metabolism in muscle, adipose tissue inflammation and neurological function. It is hypothesized that this type of exercise leads to significant improvements in insulin action and oxidative phosphorylation in muscle

ELIGIBILITY:
Inclusion criteria:

* Men and women
* Age: 30 - 65 years
* Typ-2-Diabetes (BMI > 25 kg/m²)
* Increased risk for diabetes (BMI >25 kg/m²)

Exclusion criteria:

* Acute Infection within the last 2 weeks prior to the intervention
* Autoimmune diseases and immune suppressive diseases (Leukocytes < 5000/μl)
* Intake of immunomodulating drugs (Glucocorticoids, Antihistamine, ASS)
* Pregnancy, Breastfeeding, Menstruation
* Kidney insufficiency (Creatinine > 1,5 mg/dl)
* Cardiovascular diseases
* Anemia (Hb < 12g/l), disorders of wound healing or blood clotting
* Participation in another study within the last 2 months before the investigation
* Metallic or magnetic items on or in the body
* Claustrophobia
* Thyroid dysfunction
* Intake of glitazones or insulin therapy
* Smoking (Non-smoking since > 1 year), alcohol consumption (Men > 30 g/d, Women > 20g/d) or illegal drugs
* Psychiatric disorders
* Risk for/or manifest AIDS (HIV) or Hepatitis B or C
* Night shift working
* Hypersensitivity to local anesthetics
* Cancer disease
* Lung diseases
* Systematic endurance training (>1x per week > 60min.)
* Maximal oxygen consumption (VO2 max) <20ml/min/kg
* Orthopedic disorders
* Musculoskeletal diseases

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-07; Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Improvement of Insulin sensitivity by high intensity interval training | 2 years
  High intensity interval training leads to significant improvements in insulin action and oxidative phosphorylation in skeletal muscle.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Roden, Prof., MD, Study Director — German Diabetes Center
Locations (1):
- German Diabetes Center, Düsseldorf, North Rhine-Westphalia, Germany

REFERENCES:
- [Result] Apostolopoulou M, Mastrototaro L, Hartwig S, Pesta D, Strassburger K, de Filippo E, Jelenik T, Karusheva Y, Gancheva S, Markgraf D, Herder C, Nair KS, Reichert AS, Lehr S, Mussig K, Al-Hasani H, Szendroedi J, Roden M. Metabolic responsiveness to training depends on insulin sensitivity and protein content of exosomes in insulin-resistant males. Sci Adv. 2021 Oct 8;7(41):eabi9551. doi: 10.1126/sciadv.abi9551. Epub 2021 Oct 8. PMID 34623918
- See also: Homepage — https://ddz.de/